CLINICAL TRIAL: NCT02933723
Title: Comparison of Immunogenicity of Adjuvanted and Non-Adjuvanted Influenza Vaccination in a Long-Term Care Population
Brief Title: Immunogenicity of Influenza Vaccine in Long Term Care
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Insight Therapeutics, LLC (Other)
Collaborators: Case Western Reserve University (Other); University Hospitals Cleveland Medical Center (Other); Seqirus (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: INSI-201608
Record Dates: First submitted 2016-10-10; First posted 2016-10-14 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Influenza
Keywords: influenza vaccine; nursing home; influenza; vaccination; immunity; cell-mediated immunity; humoral immunity
MeSH Terms: conditions — Influenza, Human | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blood draw- adjuvanted TIV (Experimental): individuals who received adjuvanted trivalent influenza vaccine (aTIV, Fluad) and consent to a blood draw
  Interventions: Procedure: Blood Draw
- Blood draw - nonadjuvanted TIV (Active Comparator): individuals who received nonadjuvanted trivalent influenza vaccine and consent to a blood draw
  Interventions: Procedure: Blood Draw

INTERVENTIONS:
Procedure: Blood Draw — Sampling 3 blood draws Day 0 for humoral and CMI 30 ml prior to vaccination (up to 2 week prior to vaccination) Day 7 for CMI 20 ml (+/- 1 day) Day 28 for humoral 10 ml (+/- 3 days)

SUMMARY:
The study is designed to evaluated if adjuvanted vaccine elicits higher T cell and B cell responses than non-adjuvanted standard dose influenza vaccine in nursing home residents.

DETAILED DESCRIPTION:
Summary: Study investigators will recruit residents of nursing homes that are administering a licensed influenza vaccine as their standard or care, either the trivalent influenza vaccine (Fluvirin) or the adjuvanted trivalent influenza vaccine (Fluad). Eligible residents are those or their legally authorized representatives who give written, informed consent for three blood draws over one month's time and permission to review their nursing home medical and administrative records, including information required to be submitted to Medicare including quality performance data (the Minimum Dataset or MDS) and Medicare claims data for demographic and underlying disease comparisons between our participating populations between nursing homes. The investigators propose to study up to 230 subjects in one season at a 1:1 ratio of adjuvanted vs. and non-adjuvanted vaccine.

Background: Influenza is the most common clinically important viral infection of older adults. Influenza vaccination is associated with reduced hospitalization, strokes, heart attacks and death in non-institutional older adult populations, but the benefit of influenza vaccine for the oldest population has been questioned. The adjuvanted vaccine was shown in the past to elicit higher antibody titers than non-adjuvanted TIV. This included the elderly population as well. There are far more limited data about cell-mediated immunity (CMI) and use of the adjuvanted vaccine. There are data that support that CMI is important beyond the helper function to B cells. CMI helps mitigate influenza disease if the antibodies alone are not adequately protective.

Objectives: To determine if adjuvanted vaccine elicits higher T cell and B cell responses than non-adjuvanted standard dose influenza vaccine in nursing home residents.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Medicare Certified Facility (so they have to report Minimum Data Set (MDS) data)
* Residence in a long-term care facility administering a Seqirus influenza vaccine as the standard-of-care.
* Agreed to receive the vaccine that the NH plans to give to them
* >= 65 years old
* Able to obtain consent from subject or legally authorized representative (LAR) and assent from subject
* Able to participate throughout the study period
* Resident for at least 45 days prior to enrollment

Exclusion Criteria:

* Recent illness (within 30 days) severe enough to require hospitalization or physician-directed outpatient pharmacotherapy
* Receiving chemotherapy for an active cancer

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-05-24 (Actual); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in hemagglutination inhibition (HAI) | day 0 and day 28 +/-3 days
  Fold change in antibody titers from day 0 to day 28 as determined by vaccine strain specific Hemagglutination Inhibition (HAI)
Change in microneutralization (MN) | day 0 and day 28 +/-3 days
  Fold change in antibody titers from day 0 to day 28 as determined by vaccine strain specific microneutralization

SECONDARY OUTCOMES:
Change in cell mediated immunity (CMI) - IFN-gamma | day 0 and day 7 +/-1 day
  Fold change in IFN-gamma (pg/mL) from day 0 to day 7 for vaccine strain-specific T cells
Change in cell mediated immunity (CMI) - IL-10 | day 0 and day 7 +/-1 day
  old change in IL-10 (pg/mL0 from day 0 to day 7 for vaccine strain-specific T cells

CONTACTS AND LOCATIONS:
Overall Officials: H. Edward Davidson, PharmD, Study Director — Insight Therapeutics, LLC
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nichol KL, Wuorenma J, von Sternberg T. Benefits of influenza vaccination for low-, intermediate-, and high-risk senior citizens. Arch Intern Med. 1998 Sep 14;158(16):1769-76. doi: 10.1001/archinte.158.16.1769. PMID 9738606
- [Background] Phrommintikul A, Kuanprasert S, Wongcharoen W, Kanjanavanit R, Chaiwarith R, Sukonthasarn A. Influenza vaccination reduces cardiovascular events in patients with acute coronary syndrome. Eur Heart J. 2011 Jul;32(14):1730-5. doi: 10.1093/eurheartj/ehr004. Epub 2011 Feb 2. PMID 21289042
- [Background] Frey SE, Reyes MR, Reynales H, Bermal NN, Nicolay U, Narasimhan V, Forleo-Neto E, Arora AK. Comparison of the safety and immunogenicity of an MF59(R)-adjuvanted with a non-adjuvanted seasonal influenza vaccine in elderly subjects. Vaccine. 2014 Sep 3;32(39):5027-34. doi: 10.1016/j.vaccine.2014.07.013. Epub 2014 Jul 18. PMID 25045825
- [Background] Van Buynder PG, Konrad S, Van Buynder JL, Brodkin E, Krajden M, Ramler G, Bigham M. The comparative effectiveness of adjuvanted and unadjuvanted trivalent inactivated influenza vaccine (TIV) in the elderly. Vaccine. 2013 Dec 9;31(51):6122-8. doi: 10.1016/j.vaccine.2013.07.059. Epub 2013 Aug 6. PMID 23933368
- [Background] Squarcione S, Sgricia S, Biasio LR, Perinetti E. Comparison of the reactogenicity and immunogenicity of a split and a subunit-adjuvanted influenza vaccine in elderly subjects. Vaccine. 2003 Mar 7;21(11-12):1268-74. doi: 10.1016/s0264-410x(02)00401-2. PMID 12559808
- [Background] Ansaldi F, Bacilieri S, Durando P, Sticchi L, Valle L, Montomoli E, Icardi G, Gasparini R, Crovari P. Cross-protection by MF59-adjuvanted influenza vaccine: neutralizing and haemagglutination-inhibiting antibody activity against A(H3N2) drifted influenza viruses. Vaccine. 2008 Mar 17;26(12):1525-9. doi: 10.1016/j.vaccine.2008.01.019. Epub 2008 Feb 1. PMID 18294741
- [Background] Ansaldi F, Zancolli M, Durando P, Montomoli E, Sticchi L, Del Giudice G, Icardi G. Antibody response against heterogeneous circulating influenza virus strains elicited by MF59- and non-adjuvanted vaccines during seasons with good or partial matching between vaccine strain and clinical isolates. Vaccine. 2010 Jun 7;28(25):4123-9. doi: 10.1016/j.vaccine.2010.04.030. Epub 2010 Apr 28. PMID 20433807
- [Background] Della Cioppa G, Nicolay U, Lindert K, Leroux-Roels G, Clement F, Castellino F, Galli G, Groth N, Del Giudice G. Superior immunogenicity of seasonal influenza vaccines containing full dose of MF59 ((R)) adjuvant: results from a dose-finding clinical trial in older adults. Hum Vaccin Immunother. 2012 Feb;8(2):216-27. doi: 10.4161/hv.18445. Epub 2012 Feb 1. PMID 22426371
- [Background] Wilkinson TM, Li CK, Chui CS, Huang AK, Perkins M, Liebner JC, Lambkin-Williams R, Gilbert A, Oxford J, Nicholas B, Staples KJ, Dong T, Douek DC, McMichael AJ, Xu XN. Preexisting influenza-specific CD4+ T cells correlate with disease protection against influenza challenge in humans. Nat Med. 2012 Jan 29;18(2):274-80. doi: 10.1038/nm.2612. PMID 22286307
- [Background] McElhaney JE, Xie D, Hager WD, Barry MB, Wang Y, Kleppinger A, Ewen C, Kane KP, Bleackley RC. T cell responses are better correlates of vaccine protection in the elderly. J Immunol. 2006 May 15;176(10):6333-9. doi: 10.4049/jimmunol.176.10.6333. PMID 16670345